CLINICAL TRIAL: NCT02748213
Title: An Open-Label, Randomized Phase II Study of Herceptin (Trastuzumab), Taxotere (Docetaxel), and Xeloda (Capecitabine) in Combination, Versus Herceptin (Trastuzumab) Plus Taxotere (Docetaxel), in Patients With Advanced and/or Metastatic Breast Cancers That Overexpress HER2
Brief Title: A Study of Herceptin (Trastuzumab) in Women With Human Epidermal Growth Factor Receptor (HER) 2-Positive Advanced and/or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO16419
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel; Trastuzumab

ARMS (2):
- Herceptin + Taxotere (Experimental): Participants will receive dual therapy with Herceptin and Taxotere until disease progression, unmanageable toxicity, or withdrawal.
  Interventions: Drug: Taxotere; Drug: Herceptin
- Herceptin + Taxotere + Xeloda (Experimental): Participants will receive triple therapy with Herceptin, Taxotere, and Xeloda until disease progression, unmanageable toxicity, or withdrawal.
  Interventions: Drug: Xeloda; Drug: Taxotere; Drug: Herceptin

INTERVENTIONS:
Drug: Xeloda — Participants will receive oral Xeloda, 950 mg/m^2 twice a day on Days 1 to 14 of each 21-day cycle.
  Other Names: capecitabine
  Arms: Herceptin + Taxotere + Xeloda
Drug: Taxotere — Participants will receive Taxotere, 75 milligrams per meter-squared (mg/m^2) in the Herceptin + Taxotere + Xeloda arm or 100 mg/m^2 in the Herceptin + Taxotere arm, via IV infusion on Day 1 of each 21-day cycle. The lower starting dose will be used in the triple-therapy arm.
  Other Names: docetaxel
Drug: Herceptin — Participants will receive Herceptin, 6 milligrams per kilogram (mg/kg) via IV infusion, on Day 1 of each 21-day cycle. The first dose will be a loading dose of 8 mg/kg in Cycle 1; the dose of 6 mg/kg will be given from Cycle 2 onward.
  Other Names: trastuzumab

SUMMARY:
This study will assess the efficacy and safety of intravenous (IV) trastuzumab (Herceptin) and IV docetaxel (Taxotere), with or without oral capecitabine (Xeloda), in women with previously untreated HER2-positive advanced and/or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, HER2-positive advanced and/or metastatic breast cancer not amenable to curative therapy
* At least one measurable lesion according to RECIST
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Baseline left ventricular ejection fraction (LVEF) at least 50%

Exclusion Criteria:

* Pregnant, lactating, or women of childbearing potential who are not surgically sterile or not willing to use adequate contraceptive methods
* Previous treatment with Herceptin or other anti-HER therapies, or any previous chemotherapy for advanced or metastatic disease
* Past medical history significant for any cardiac or central nervous system (CNS) disorders
* Poor hematologic, renal, or hepatic function
* Chronic corticosteroid therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2002-02; Primary Completion 2006-03 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (49):
- Australia (7):
  - Adelaide
  - Brisbane
  - Camperdown
  - Geelong
  - Melbourne
  - Perth
  - Southport
- Brazil (3):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (3):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Québec, Quebec
- San José, Costa Rica
- Turku, Finland
- France (6):
  - Besançon
  - Grenoble
  - Marseille
  - Paris
  - Pierre-Bénite
  - Rennes
- Greece (3):
  - Athens
  - Heraklion
  - Pátrai
- Guatemala City, Guatemala
- Italy (5):
  - Legnago
  - Noale
  - Rozzano
  - Trento
  - Treviglio
- Mexico (3):
  - Distrito Federal
  - Mérida
  - Monterrey
- Panama City, Panama
- Poland (2):
  - Gdansk
  - Szczecin
- Spain (4):
  - Barcelona
  - Lleida
  - Sabadell, Barcelona
  - Zaragoza
- Sweden (2):
  - Karlstad
  - Västerås
- United Kingdom (7):
  - Ipswich
  - Leeds
  - Manchester
  - Northwood
  - Oxford
  - Southampton
  - Weston-super-Mare

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241

RESULTS

PARTICIPANT FLOW:
Groups:
- Herceptin + Taxotere + Xeloda: Participants received triple therapy with Herceptin, Taxotere, and Xeloda until disease progression, unmanageable toxicity, or withdrawal. Herceptin and Taxotere were given via intravenous (IV) infusion on Day 1 of each 21-day cycle. The first dose of Herceptin was a loading dose of 8 milligrams per kilogram (mg/kg) in Cycle 1, and a maintenance dose of 6 mg/kg was given from Cycle 2 through the end of treatment. The dose of Taxotere was 75 milligrams per meter-squared (mg/m^2), with adjustments allowed only for toxicity. Xeloda was given orally as 950 mg/m^2 twice a day on Days 1 to 14 of each 21-day cycle, with adjustments allowed only for toxicity.
- Herceptin + Taxotere: Participants received dual therapy with Herceptin and Taxotere until disease progression, unmanageable toxicity, or withdrawal. Treatments were given via IV infusion on Day 1 of each 21-day cycle. The first dose of Herceptin was a loading dose of 8 mg/kg in Cycle 1, and a maintenance dose of 6 mg/kg was given from Cycle 2 through the end of treatment. The dose of Taxotere was 100 mg/m^2, with adjustments allowed only for toxicity.
Period: Overall Study
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Started | 113 | 112
Treated | 112 | 110
Completed | 0 (*The reason "Refused Treatment" also includes those who did not cooperate or withdrew consent.) | 0
Not Completed | 113 | 112
Not completed — Withdrawal Prior to Treatment | 1 | 2
Not completed — Abnormal Laboratory Test | 1 | 0
Not completed — Adverse Event or Intercurrent Illness | 5 | 11
Not completed — Death | 5 | 3
Not completed — Insufficient Therapeutic Response | 56 | 57
Not completed — Violation of Selection Criteria | 2 | 0
Not completed — Protocol Violation | 6 | 4
Not completed — Refused Treatment* | 6 | 6
Not completed — Failure to Return | 1 | 0
Not completed — Other | 30 | 29

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) Population: All participants, according to randomization scheme, who received at least one dose of study medication.
Groups:
- Herceptin + Taxotere + Xeloda: Participants received triple therapy with Herceptin, Taxotere, and Xeloda until disease progression, unmanageable toxicity, or withdrawal. Herceptin and Taxotere were given via IV infusion on Day 1 of each 21-day cycle. The first dose of Herceptin was a loading dose of 8 mg/kg in Cycle 1, and a maintenance dose of 6 mg/kg was given from Cycle 2 through the end of treatment. The dose of Taxotere was 75 mg/m^2, with adjustments allowed only for toxicity. Xeloda was given orally as 950 mg/m^2 twice a day on Days 1 to 14 of each 21-day cycle, with adjustments allowed only for toxicity.
- Total: Total of all reporting groups
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere | Total
Number analyzed (Participants) | 112 | 110 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (11.18) | 51.6 (10.74) | 52.1 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 110 | 222
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Tumor response was assessed by RECIST during the study. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels. PR was defined as greater than or equal to (≥) 30 percent (%) decrease in sum of longest diameter (LD) of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥4 weeks after the initial assessment of CR or PR. The percentage of participants with a best overall response for CR or PR was reported. The exact 95% confidence interval (CI) for one-sample binomial was determined using the Pearson-Clopper method.
Time Frame: Tumor assessments at Baseline, then every 6 weeks until Cycle 8 (cycle length of 21 days), then every 12 weeks until progressive disease and/or one year after enrollment; thereafter according to routine clinical practice (up to 66 months overall)
Population: Full Analysis Set (FAS) Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Number analyzed (Participants) | 112 | 110
percentage of participants | 70.5 [61.18 to 78.77] | 72.7 [63.41 to 80.78]
Statistical Analysis 1: Comparison: Herceptin + Taxotere + Xeloda vs Herceptin + Taxotere; Test type: Superiority or Other; p = 0.717, Chi-squared; Difference in Response Rates = 2.2, 95% CI 2-sided [-10.17 to 14.56] — The approximate 95% CI for the difference in response (CR or PR) rates was determined using the Hauck-Anderson correction

2. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to RECIST
Description: Tumor response was assessed by RECIST during the study. Disease progression or progressive disease (PD) was defined as ≥20% increase in sum LD in reference to the smallest on-treatment sum LD, or the appearance of new lesions. The percentage of participants who died or experienced PD was reported.
Time Frame: as for outcome 1
Population: FAS Population.
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Number analyzed (Participants) | 112 | 110
percentage of participants | 67.9 | 77.3

3. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST
Description: Tumor response was assessed by RECIST during the study. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-treatment sum LD, or the appearance of new lesions. PFS was defined as the time from start of treatment to the first event of death or PD. Participants without event at the time of analysis were censored at the latest date of last tumor assessment or last date in drug log. The median duration of PFS and corresponding 95% CI were estimated by Kaplan-Meier analysis and expressed in months.
Time Frame: as for outcome 1
Population: FAS Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Number analyzed (Participants) | 112 | 110
months | 17.9 [14 to 21] | 12.8 [10 to 16]
Statistical Analysis 1: Comparison: Herceptin + Taxotere + Xeloda vs Herceptin + Taxotere; Test type: Superiority or Other; p = 0.0449, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.53 to 0.99] — Hazard Ratio (HR) calculated using Herceptin + Taxotere arm as reference

4. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants who died from any cause was reported.
Time Frame: Continuously during treatment (up to 66 months) and at any time after treatment discontinuation until 18 months after last participant enrolled (up to 66 months overall)
Population: FAS Population.
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Number analyzed (Participants) | 112 | 110
percentage of participants | 35.7 | 41.8

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start of treatment to date of death for any reason. Participants who were alive at the time of analysis were censored at the latest date of last tumor assessment, last drug intake, or last follow-up information. The median duration of OS and corresponding 95% CI were estimated by Kaplan-Meier analysis and expressed in months.
Time Frame: as for outcome 4
Population: FAS Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Number analyzed (Participants) | 112 | 110
months | 43.5 [40 to 50] | 47.3 [32 to NA] — The upper limit of the 95% CI was not reached due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Herceptin + Taxotere + Xeloda vs Herceptin + Taxotere; Test type: Superiority or Other; p = 0.4758, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.56 to 1.32] — HR calculated using Herceptin + Taxotere arm as reference

6. Secondary Outcome: Duration of Response (DOR) According to RECIST
Description: Tumor response was assessed by RECIST during the study. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels. PR was defined as ≥30% decrease in sum LD of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥4 weeks after the initial assessment of CR or PR. DOR was defined as the time from first assessment of CR or PR until the first occurrence of documented PD, death, or withdrawal. The median DOR was reported and expressed in months.
Time Frame: as for outcome 1
Population: FAS Population. The "Number of Participants Analyzed" reflects the number of participants with a best overall response of CR or PR who provided evaluable data for the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Number analyzed (Participants) | 78 | 80
months | 15.9 [2.4 to 64.7] | 13.4 [2.1 to 55.1]

ADVERSE EVENTS:
Time Frame: Continuously during treatment (up to 66 months) and up to 28 days after last dose (up to 66 months overall)
Description: Safety Population: All randomized participants, according to treatment actually received, who received at least one dose of study medication.
Arm/Group | Herceptin + Taxotere + Xeloda | Herceptin + Taxotere
Serious Adverse Events (participants affected / at risk) | 52/112 | 51/110
Other Adverse Events (participants affected / at risk) | 112/112 | 107/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin + Taxotere + Xeloda (N=112) | Herceptin + Taxotere (N=110)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 26
Neutropenia (Blood and lymphatic system disorders) | 7 | 7
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 5 | 1
Bronchopneumonia (Infections and infestations) | 3 | 0
Central line infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 3 | 4
Oedema peripheral (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Inflammation of wound (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Pitting oedema (General disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 3
Diplegia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurosis (Psychiatric disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin + Taxotere + Xeloda (N=112) | Herceptin + Taxotere (N=110)
Diarrhoea (Gastrointestinal disorders) | 75 | 55
Nausea (Gastrointestinal disorders) | 61 | 39
Vomiting (Gastrointestinal disorders) | 37 | 30
Constipation (Gastrointestinal disorders) | 29 | 23
Stomatitis (Gastrointestinal disorders) | 29 | 19
Abdominal pain (Gastrointestinal disorders) | 25 | 16
Dyspepsia (Gastrointestinal disorders) | 22 | 12
Abdominal pain upper (Gastrointestinal disorders) | 13 | 5
Gastritis (Gastrointestinal disorders) | 6 | 4
Haemorrhoids (Gastrointestinal disorders) | 8 | 1
Odynophagia (Gastrointestinal disorders) | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 76 | 68
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 57 | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 28 | 20
Rash (Skin and subcutaneous tissue disorders) | 22 | 18
Onycholysis (Skin and subcutaneous tissue disorders) | 20 | 14
Erythema (Skin and subcutaneous tissue disorders) | 13 | 10
Skin reaction (Skin and subcutaneous tissue disorders) | 15 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 10 | 3
Nail toxicity (Skin and subcutaneous tissue disorders) | 4 | 6
Onychomadesis (Skin and subcutaneous tissue disorders) | 6 | 2
Asthenia (General disorders) | 35 | 35
Oedema peripheral (General disorders) | 28 | 42
Fatigue (General disorders) | 35 | 29
Mucosal inflammation (General disorders) | 34 | 30
Pyrexia (General disorders) | 25 | 19
Chest pain (General disorders) | 9 | 10
Chills (General disorders) | 10 | 9
Oedema (General disorders) | 3 | 15
Pain (General disorders) | 6 | 8
Headache (Nervous system disorders) | 20 | 28
Paraesthesia (Nervous system disorders) | 11 | 20
Dizziness (Nervous system disorders) | 12 | 16
Dysgeusia (Nervous system disorders) | 17 | 11
Neuropathy peripheral (Nervous system disorders) | 13 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 13
Neuropathy (Nervous system disorders) | 11 | 11
Lethargy (Nervous system disorders) | 8 | 13
Neurotoxicity (Nervous system disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 28
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 38
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 11
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 19
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Neutropenia (Blood and lymphatic system disorders) | 35 | 23
Anaemia (Blood and lymphatic system disorders) | 15 | 19
Leukopenia (Blood and lymphatic system disorders) | 10 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 6
Lacrimation increased (Eye disorders) | 25 | 22
Conjunctivitis (Eye disorders) | 15 | 14
Dry eye (Eye disorders) | 7 | 7
Vision blurred (Eye disorders) | 3 | 6
Nasopharyngitis (Infections and infestations) | 15 | 12
Rhinitis (Infections and infestations) | 13 | 11
Influenza (Infections and infestations) | 13 | 10
Urinary tract infection (Infections and infestations) | 8 | 11
Hot flush (Vascular disorders) | 9 | 14
Lymphoedema (Vascular disorders) | 8 | 13
Phlebitis (Vascular disorders) | 6 | 4
Anorexia (Metabolism and nutrition disorders) | 23 | 19
Insomnia (Psychiatric disorders) | 10 | 12
Depression (Psychiatric disorders) | 4 | 10
Anxiety (Psychiatric disorders) | 4 | 8
Dysuria (Renal and urinary disorders) | 8 | 6
Weight decreased (Investigations) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.